CLINICAL TRIAL: NCT03658668
Title: Study of the Combined Effect of Transcranial Direct Current Stimulation (tDCS) and Physical Activity on Gait and Functional Mobility in Participants With Multiple Sclerosis
Brief Title: Combined Effect of Transcranial Direct Current Stimulation (tDCS) and Physical Activity on Gait and Functional Mobility in Participants With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18-00534
Record Dates: First submitted 2018-08-14; First posted 2018-09-05 (Actual); Results first posted 2023-08-16 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-07

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- active tDCS+PA (Experimental)
  Interventions: Device: active tDCS; Other: Physical Activity (PA)
- sham tDCS+PA (Sham Comparator)
  Interventions: Device: sham tDCS; Other: Physical Activity (PA)

INTERVENTIONS:
Device: active tDCS — tDCS is a therapeutic treatment that utilizes low amplitude direct currents (<4 mA) to induce changes in cortical excitability.
  Other Names: Soterix 1x1 tDCS mini-CT
  Arms: active tDCS+PA
Device: sham tDCS — During a sham session, the device is programmed to ramp up to the desired intensity (target 2.5 mA) and ramp down for the initial 60 seconds, with no current delivery during the session, and then again at the end of the session. These brief periods of stimulation serve to mimic the effects of a true stimulation session.
  Arms: sham tDCS+PA
Other: Physical Activity (PA) — 20 minutes of cycling on an ergonomic cross-trainer

SUMMARY:
This study is aimed to test the efficacy of transcranial direct current stimulation (tDCS) combined with a physical activity (PA) program, in 80 individuals affected by Multiple Sclerosis (MS). In particular, this study will evaluate the efficacy of tDCS when administered simultaneously with PA on walking, functional mobility, and fatigue.

The subjects enrolled will be randomly assigned to the active group (active tDCS+PA) or the sham group (sham tDCS+PA).

Portions of this study may be completed remotely.

ELIGIBILITY:
Inclusion Criteria:

* Stable and continuous access to internet service at home
* Adequate home facilities (enough space, access to quiet and distraction free area)
* Definite MS diagnosis, subtype relapsing-remitting (RR-MS)
* Disability Status Scale (EDSS) from 1 to 6.5 with clinically significant gait deviations
* Clinically stable and stable on treatment with disease modifying agents at least from 6 months
* Able to independently walk with or without an assisting device (i.e. cane, crutches or walking frames) for medium-long distance
* Absence of other associated medical conditions that would prevent participants from performing physical activity, such as cardiorespiratory and severe osteoarticular disorders
* Able to use study equipment
* Able to commit 10 consecutive daily sessions of tDCS while performing physical program with baseline and follow-up visits
* Able to understand the informed consent process and provide consent to participate in the study

Exclusion Criteria:

* Visual, auditory and motor deficits that would prevent full ability to understand study, as judged by treating neurologist or study staff
* Primary psychiatric disorder that would influence ability to participate
* Receiving current treatment for epilepsy
* Uncontrolled headaches and migraines. In addition, if a subject has had a change in the rate or severity of head pressure, headache, or migraine in the past two weeks, they are excluded
* History of head trauma (e.g., head injury, brain surgery) or medical device implanted in the head (such as Deep Brain Stimulator) or in the neck (such as a Vagus Nerve Stimulator)
* Any skin disorder/sensitive skin (e.g., eczema, severe rashes), blisters, open wounds, burn including sunburns, cuts or irritation, or other skin defects which compromise the integrity of the skin at or near stimulation locations (where electrodes are placed)
* Treatment for a communicable skin disorder currently or over the past 12 months
* History of uncontrolled or labile hypertension
* Other serious uncontrolled medical condition (e.g. cancer or acute myocardial infarction)
* Wide Range Achievement Test-4th Edition (WRAT-4) Reading Recognition score < 85
* History of clinically significant abnormalities on electrocardiogram (EKG)
* Presence of chronic medical illness and/or severe ataxia
* Botulinum toxin injection within the past 4 months or functional surgery in the past 6 months
* Alcohol or other substance use disorder
* Pregnant or breastfeeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-10-03 (Actual); Primary Completion 2021-06-10 (Actual); Study Completion 2021-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leigh Charvet, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

REFERENCES:
- [Derived] Pilloni G, Choi C, Coghe G, Cocco E, Krupp LB, Pau M, Charvet LE. Gait and Functional Mobility in Multiple Sclerosis: Immediate Effects of Transcranial Direct Current Stimulation (tDCS) Paired With Aerobic Exercise. Front Neurol. 2020 May 5;11:310. doi: 10.3389/fneur.2020.00310. eCollection 2020. PMID 32431658

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active tDCS+PA | Sham tDCS+PA
Started | 13 | 9
Completed | 12 | 8
Not Completed | 1 | 1
Not completed — Time Commitment | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active tDCS+PA | Sham tDCS+PA | Total
Number analyzed (Participants) | 12 | 8 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.4 (12.3) | 55 (7.55) | 54.3 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 4 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 1 | 11
  Not Hispanic or Latino | 1 | 7 | 8
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 8 | 6 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 12 | 8 | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in Gait Velocity
Description: Measured by a 10 meter walk test using wearable inertial sensors
Time Frame: Baseline, Follow-Up Visit (3 days after final treatment session, up to 4 weeks)
Measure: Mean (Standard Deviation); unit: meters/second (m/s)
Arm/Group | Active tDCS+PA | Sham tDCS+PA
Number analyzed (Participants) | 9 | 6
meters/second (m/s) | 0.33 (0.32) | 0.01 (0.33)

2. Primary Outcome: Change in Stride Length
Description: Measured by a 10 meter walk test using wearable inertial sensors
Time Frame: Baseline, Follow-Up Visit (3 days after final treatment session, up to 4 weeks)
Measure: Mean (Standard Deviation); unit: meters (m)
Arm/Group | Active tDCS+PA | Sham tDCS+PA
Number analyzed (Participants) | 9 | 6
meters (m) | 0.32 (0.17) | -0.02 (0.2)

3. Secondary Outcome: Percent of tDCS Sessions Completed
Time Frame: End of Final Treatment Session (Up to Week 3)
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Active tDCS+PA | Sham tDCS+PA
Number analyzed (Participants) | 9 | 6
Percentage | 100 (0) | 100 (0)

4. Secondary Outcome: Change in 12-item Multiple Sclerosis Walking Scale Score
Description: 12-item questionnaire assessing how multiple sclerosis (MS) affects walking abilities. Items are ranked on a scale from 1 (not at all) to 5 (extremely). The total score is the sum of responses and ranges from 12 to 60; higher scores indicate greater impact of MS on walking abilities.
Time Frame: Baseline, Follow-Up Visit (3 days after final treatment session, up to 4 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active tDCS+PA | Sham tDCS+PA
Number analyzed (Participants) | 9 | 6
score on a scale | -4.9 (3.2) | -2.5 (2.9)

5. Secondary Outcome: Change 21-item Modified Fatigue Impact Scale Score
Description: 21-item questionnaire assessing how fatigue may affect a person. Items are ranked on a scale from 0 (never) to 4 (almost always). The total score is the sum of responses and ranges from 0 to 84; scores indicate greater impact of fatigue.
Time Frame: Baseline, Follow-Up Visit (3 days after final treatment session, up to 4 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active tDCS+PA | Sham tDCS+PA
Number analyzed (Participants) | 9 | 6
score on a scale | -12.4 (10.4) | 1.6 (8.7)

ADVERSE EVENTS:
Time Frame: 10 days
Description: Standard questionnaire.
Arm/Group | Active tDCS+PA | Sham tDCS+PA
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/9
Other Adverse Events (participants affected / at risk) | 12/13 | 9/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active tDCS+PA (N=13) | Sham tDCS+PA (N=9)
Tingling at the electrode site (General disorders) | 10 | 8
Itching at the electrode site (General disorders) | 9 | 6
Warmth Sensation at the electrode site (General disorders) | 5 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-09): https://cdn.clinicaltrials.gov/large-docs/68/NCT03658668/Prot_SAP_000.pdf